CLINICAL TRIAL: NCT02535143
Title: The Impact of Energy Drinks on the Manual Dexterity of Final Year Dental Students
Brief Title: Impact of Energy Drinks on the Manual Dexterity of Final Year Dental Students
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Dr Sharat Pani, Assistant Professor, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: FUGRP/2014/183.
Record Dates: First submitted 2015-08-26; First posted 2015-08-28 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Hand Skill, Relative
MeSH Terms: interventions — Taurine; Energy Drinks

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test Group (Experimental): Group will prepare a test cavity in an acrylic block. They will receive 250 ml of a commercially available energy drink containing caffeine and taurine (Red Bull, Red Bull GmBh Austria) three hours after the last meal. The participants will then be required to perform a post intervention test cavity preparation 30 minutes after consuming the drink.
  Interventions: Other: Test Cavity Preparation; Drug: Taurine; Other: Post intervention test cavity
- Control Group (Placebo Comparator): Group will prepare a test cavity in an acrylic block. They will receive 250ml of a commercially available carbonated apple juice (Appy Fizz, Parle Agro, Mumbai, India) three hours after the last meal. The participants will then be required to perform a post intervention test cavity preparation 30 minutes after consuming the drink.
  Interventions: Other: Test Cavity Preparation; Other: Post intervention test cavity; Dietary Supplement: Carbonated Apple Juice

INTERVENTIONS:
Other: Test Cavity Preparation — Subjects will be asked to prepare a cavity 2mmx 2mmx 2mm in an acrylic block using an airotor and a tungsten carbide bur prior to consuming the test drink
  Other Names: Dexterity test
Drug: Taurine — 250 ml of commercially available taurine containing energy drink to be administered three hours after the last meal and half an hour prior to performing the second test cavity
  Other Names: Energy Drink
  Arms: Test Group
Other: Post intervention test cavity — Subjects will be asked to prepare a cavity 2mmx 2mmx 2mm in an acrylic block 30 minutes after consuming the intervention drink using an airotor and a tungsten carbide bur prior to consuming the test drink
Dietary Supplement: Carbonated Apple Juice — 250ml of commercially available carbonated apple juice to be administered three hours after the last meal and half an hour prior to performing the second test cavity
  Other Names: Appy FIzz (Parle Agro, India)
  Arms: Control Group

SUMMARY:
This study aims to test the hypothesis that there was a relationship between the consumption of energy drinks and the manual dexterity skills of final year dental students.

Identification of baseline caffeine consumption and selection of sample Baseline caffeine consumption will be identified by distributing the caffeine consumption questionnaire to all the final year students of the Riyadh Colleges of Dentistry and Pharmacy. The study will recruit 60 students who are moderate caffeine consumers. To avoid the confounding effect of nicotine consumption, the study will only recruit non-smokers .female candidates taken oral contraceptives and Subjects with any history of renal disease will be excluded.

All subjects will be required to prepare a box 2mmx2mmx2mm using a high speed handpiece (NSK, Japan) and a no.330 cutting bur. Each participant will be allowed two attempts to cut the cavity in each test both cavities will be selected for assessment. The ability of the participants to reproduce the dimensions (2mmx2mmx2mm) and the time taken to complete the task will be used as criteria to evaluate dexterity. The participants will be required to perform the test before and 30 minutes after energy drink exposure.

Energy Drink Exposure Subjects will be given 330ml of an energy three hours after the last meal in the other hand the control group will be receiving a placebo drink .

Dexterity outcomes will be compared before and after exposure to the energy drink using the paired t test. Outcomes will be compared between different groups and different time intervals using the two way, multiple measures ANOVA. All data will be analyzed using the SPSS ver.21 data processing software.

DETAILED DESCRIPTION:
The dentistry training program has been reported to be a stressful one; and while academic pressures are high, the high level of dexterity skills that dentistry demands are often cited as a major source of stress. There is some research on the impact that caffeine in general and energy drinks in particular can have on academic performance, however, there is considerably less data on the impact of these drinks on manual dexterity. This study aims to test the hypothesis that there was a relationship between the consumption of energy drinks and the manual dexterity skills of final year dental students.

Identification of baseline caffeine consumption and selection of sample Baseline caffeine consumption will be identified by distributing the caffeine consumption questionnaire to all the final year students of the Riyadh Colleges of Dentistry and Pharmacy. Based on the caffeine consumption score the study will recruit 60 moderate. To avoid the confounding effect of nicotine consumption, the study will only recruit non-smokers .female candidates taken oral contraceptives will be eliminated due to the correlation between them and caffeine. Subjects with any history of renal disease will be prevented from participation in the study Test for manual dexterity Acrylic blocks (2cmx2cmx2cm) will be prepared using a standardized mold. All subjects will be required to prepare a box 2mmx2mmx2mm using a high speed handpiece (NSK, Japan) and a no.330 cutting bur. Each participant will be allowed two attempts to cut the cavity in each test both cavities will be selected for assessment. The ability of the participants to reproduce the dimensions (2mmx2mmx2mm) and the time taken to complete the task will be used as criteria to evaluate dexterity. The participants will be required to perform the test before and 30 minutes after energy drink exposure.

Energy Drink Exposure Subjects in the test group (n 30) will be given 330ml of an energy drink containing caffeine, sugar and taurine (Red Bull, Red Bull GmbH, Austria Vienna) three hours after the last meal in the other hand the control group (n30) will be receiving a placebo drink which is apple juice.

Statistical Analysis Dexterity outcomes will be compared before and after exposure to the energy drink using the paired t test. Outcomes will be compared between different groups and different time intervals using the two way, multiple measures ANOVA. All data will be analyzed using the SPSS ver.21 data processing software.

ELIGIBILITY:
Inclusion Criteria:

* Final year dental student
* Able to prepare acceptable test cavity (2mmx2mmx2mm) prior to intervention

Exclusion Criteria:

* Smokers
* Women on Oral Contraceptives
* History of Renal Disease

Ages: 21 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Cavity Accuracy in mm | Immediate
  Accuracy of the test cavity prepared in mm

SECONDARY OUTCOMES:
Time taken to prepare the cavity in seconds | immediate
  Time taken in seconds to prepare the test cavity

CONTACTS AND LOCATIONS:
Overall Officials: Hezekiah A Mosadomi, DMD, Study Chair — Riyadh Colleges of Dentistry and Pharmacy
Locations (1):
- Riyadh Colleges of Dentistry and Pharmacy, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almalak H, Albluwi AI, Alkhelb DA, Alsaleh HM, Khan TM, Hassali MA, Aljadhey H. Students' attitude toward use of over the counter medicines during exams in Saudi Arabia. Saudi Pharm J. 2014 Apr;22(2):107-12. doi: 10.1016/j.jsps.2013.02.004. Epub 2013 Mar 21. PMID 24648821
- [Background] Alsunni AA, Badar A. Energy drinks consumption pattern, perceived benefits and associated adverse effects amongst students of University of Dammam, Saudi Arabia. J Ayub Med Coll Abbottabad. 2011 Jul-Sep;23(3):3-9. PMID 23272423
- [Background] Arai YC, Kandatsu N, Ito H, Sato Y, Satake Y, Mizutani M, Ushida T, Komatsu T. Induction and emergence behavior of children undergoing general anesthesia correlates with maternal salivary amylase activity before the anesthesia. Acta Anaesthesiol Scand. 2008 Feb;52(2):285-8. doi: 10.1111/j.1399-6576.2007.01527.x. Epub 2007 Nov 14. PMID 18005374
- [Background] Arria AM, Bugbee BA, Caldeira KM, Vincent KB. Evidence and knowledge gaps for the association between energy drink use and high-risk behaviors among adolescents and young adults. Nutr Rev. 2014 Oct;72 Suppl 1(0 1):87-97. doi: 10.1111/nure.12129. PMID 25293548
- [Background] Azagba S, Langille D, Asbridge M. An emerging adolescent health risk: caffeinated energy drink consumption patterns among high school students. Prev Med. 2014 May;62:54-9. doi: 10.1016/j.ypmed.2014.01.019. Epub 2014 Feb 4. PMID 24502849
- [Background] GOLDBERG AA, JEFFERIES HS. Potentiation of insulin hypoglycaemia by nicotinyl taurine (beta-nicotinamidoethanesulphonic acid). Q J Pharm Pharmacol. 1946 Jan-Mar;19:48-53. No abstract available. PMID 20982931
- [Background] Pai KM, Kamath A, Goel V. Effect of Red Bull energy drink on muscle performance: an electromyographic overview. J Sports Med Phys Fitness. 2015 Dec;55(12):1459-65. Epub 2014 Oct 21. PMID 25331270
- [Background] Spierer DK, Blanding N, Santella A. Energy drink consumption and associated health behaviors among university students in an urban setting. J Community Health. 2014 Feb;39(1):132-8. doi: 10.1007/s10900-013-9749-y. PMID 23959655